CLINICAL TRIAL: NCT01456559
Title: Non-invasive Detection of Mild Hypovolemia Using Pleth Variability Index (PVI) During Spontaneous Breathing
Brief Title: Detection of Hypovolemia Using Pleth Variability Index (PVI)
Status: Completed | Type: Observational
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Lena Nilsson, MD, PhD, University Hospital, Linkoeping
Other Study IDs: Vers 2011-07-11
Record Dates: First submitted 2011-10-16; First posted 2011-10-20 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Hypovolemia
Keywords: Hypovolemia; Lower body negative pressure; Photoplethysmography
MeSH Terms: conditions — Hypovolemia | interventions — Lower Body Negative Pressure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Lower body negative pressure (LBNP) — The purpose with the planned study is to study pleth variability index (PVI) as a non invasive indicator for mild hypovolemia during spontaneous breathing in healthy subjects. Lower body negative pressure (LBNP), a well established technique, is used to create defined levels of hypovolemia.
  Baseline data are recorded with the subjects in the supine position breathing with normal tidal volume without PEEP and without LBNP applied. Data are then recorded with LBNP applied in two steps (40 and 15 mmHg). Recordings are continued 5 minutes after releasing the negative pressure. Data are collected in total in four different series; normal tidal volume without PEEP; normal tidal volume with PEEP 5cm H2O; three doubled tidal volume without PEEP; three doubled tidal volume with PEEP 5 cm H20.

SUMMARY:
The purpose with the planned study is to study Pleth Variability Index (PVI) as a non invasive indicator for mild hypovolemia during spontaneous breathing in healthy subjects. Lower body negative pressure (LBNP), a well established technique is used to create defined levels of hypovolemia.

Primary hypothesis: By applying a breathing resistance (positive end expiratory pressure PEEP) to spontaneous breathing, the respiratory synchronous variation in the pulse oximeter signal (PVI) is enhanced and enables PVI to detect and grade the level of mild hypovolemia.

Secondary hypothesis: 1) When tidal volume is increased, the respiratory synchronous variation in the pulse oximeter signal (PVI) will also increase. 2) The earlobe is superior to the finger in detecting PVI 3) Hemoglobin (Hb), detected non invasively by pulse oximetry, is not affected by hypovolemia created by LBNP

DETAILED DESCRIPTION:
The subjects are placed supine on a bed. Non invasive equipment for recording pulse and blood pressure is placed on a finger on the right hand. From this equipment total peripheral resistance and cardiac output are recorded. A pulse oximeter for saturation, perfusion index and PVI is placed on a finger and on the ear lobe. Data are recorded in parallel from the finger and the ear lobe. In addition non invasive haemoglobin (Hb) is recorded from the pulse oximeter on the finger. The subjects breathe through a mask connected to a simple Y-connector with an inspiratory valve on one side and an expiratory valve on the other. A positive pressure valve is applied on the expiratory side. Tidal volume is measured on-line by a connector connected to a spirometer and the tidal volume is displayed to the subjects. Stroke volume, total peripheral resistance and cardiac output is measured using ultra sound via the jugular fossa.

Baseline data are recorded with the subjects in the supine position breathing with normal tidal volume without PEEP and without LBNP applied. Data are then recorded with LBNP applied in two steps (40 and 15 mmHg). Recordings are continued 5 minutes after releasing the negative pressure. Data are collected in total in four different series; normal tidal volume without PEEP; normal tidal volume with PEEP 5cm H2O; three doubled tidal volume without PEEP; three doubled tidal volume with PEEP 5 cm H20. Respiratory rate is not controlled. The order of the four series is randomized. Between the series a 20 minute period of rest is allowed to the subjects. This period is also necessary to restore steady state between provocations.

ELIGIBILITY:
Inclusion Criteria:

* Subjects without any heart or lung disease

Exclusion Criteria:

* Smoking
* Drugs affecting circulatory or respiratory system

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy subjects between 18-30 years old without any medications affecting circulatory or respiratory system
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pleth Variability Index (PVI) | Participants will be followed only during the experimental study, 3 hours.
  Primary endpoint: PVI at two different predefined levels of hypovolemia created by using lower negative body pressure, 40 and 15 mmHg, respectively.

SECONDARY OUTCOMES:
Pleth Variability Index (PVI) | Participants will be followed only during the experiments, for 3 hours
  Correlation between PVI as an indication of hypovolemia measured simultaneously from two locations, ear lobe and finger.
SpHb | Participants will be followed during the experiments, for 3 hours
  Non-invasive hemoglobin (SpHb) is followed during mild hypovolemia created by lower body negative pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Lena Nilsson, MD, PhD, Principal Investigator — Anestesi- och operationskliniken, Linköping Universtity Hospital, S-581 85 Linköping, Sweden
Locations (2):
- Sweden (2):
  - Universitetssjukhuset, Linköping
  - Anestesi- och operationskliniken, Universitetssjukhuset, Linköping

REFERENCES:
- [Background] Cannesson M, Desebbe O, Rosamel P, Delannoy B, Robin J, Bastien O, Lehot JJ. Pleth variability index to monitor the respiratory variations in the pulse oximeter plethysmographic waveform amplitude and predict fluid responsiveness in the operating theatre. Br J Anaesth. 2008 Aug;101(2):200-6. doi: 10.1093/bja/aen133. Epub 2008 Jun 2. PMID 18522935
- [Background] Cooke WH, Ryan KL, Convertino VA. Lower body negative pressure as a model to study progression to acute hemorrhagic shock in humans. J Appl Physiol (1985). 2004 Apr;96(4):1249-61. doi: 10.1152/japplphysiol.01155.2003. PMID 15016789
- [Background] Keller G, Cassar E, Desebbe O, Lehot JJ, Cannesson M. Ability of pleth variability index to detect hemodynamic changes induced by passive leg raising in spontaneously breathing volunteers. Crit Care. 2008;12(2):R37. doi: 10.1186/cc6822. Epub 2008 Mar 6. PMID 18325089
- [Background] Shelley KH, Jablonka DH, Awad AA, Stout RG, Rezkanna H, Silverman DG. What is the best site for measuring the effect of ventilation on the pulse oximeter waveform? Anesth Analg. 2006 Aug;103(2):372-7, table of contents. doi: 10.1213/01.ane.0000222477.67637.17. PMID 16861419
- [Background] Nilsson L, Goscinski T, Kalman S, Lindberg LG, Johansson A. Combined photoplethysmographic monitoring of respiration rate and pulse: a comparison between different measurement sites in spontaneously breathing subjects. Acta Anaesthesiol Scand. 2007 Oct;51(9):1250-7. doi: 10.1111/j.1399-6576.2007.01375.x. Epub 2007 Aug 15. PMID 17711563
- [Derived] Nilsson LM, Lindenberger DM, Hahn RG. The effect of positive end-expiratory pressure and tripled tidal volume on pleth variability index during hypovolaemia in conscious subjects: a volunteer study. Eur J Anaesthesiol. 2013 Nov;30(11):671-7. doi: 10.1097/EJA.0b013e32836394c0. PMID 23839074